CLINICAL TRIAL: NCT03251209
Title: Influence of Mental Practice on Manual Dexterity Associated Before and After Physical Practice in Patients With Stroke Sequelae
Brief Title: Mental Practice in Post-stroke Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Roberta de Oliveira Cacho, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.978.586/2017
Record Dates: First submitted 2017-08-07; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Stroke Sequelae; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Post-stroke participants receive the mental practice before the physical practice. The activities will be presented in a videotherapy way.
  Interventions: Other: Physical practice; Other: Mental practice; Other: Videotherapy
- Group 2 (Experimental): Post-stroke participants receive the mental practice after the physical practice. The activities will be presented in a videotherapy way.
  Interventions: Other: Physical practice; Other: Mental practice; Other: Videotherapy
- Group 3 (Active Comparator): Post-stroke participants receive only physical practice. The activities will be presented in a videotherapy way.
  Interventions: Other: Physical practice; Other: Videotherapy

INTERVENTIONS:
Other: Physical practice — Physical Practice: reproduce through the motor execution (4 distinct tasks: stacking cubes, opposition of fingers with precision gripping, passing water from one glass to another, sequencing of bottles), the activities assisted in the video (5 minutes / task).
Other: Mental practice — Mental practice: think about the tasks watched in the videotherapy (4 distinct tasks: stacking cubes, opposition of fingers with precision gripping, passing water from one glass to another, sequencing of bottles) for 5 minutes / task.
  Arms: Group 1; Group 2
Other: Videotherapy — Videotherapy, being 2 minutes per task (4 distinct tasks: stacking cubes, opposition of fingers with precision gripping, passing water from one glass to another, sequencing of bottles)

SUMMARY:
Among the limitations caused by cerebrovascular accident (CVA), the upper limb (MS) undergoes changes that limit the individual in his ability to maintain an active social life. Mental Practice (MP) consists of the internal reproduction of an event, which is repeated extensively in order to learn or improve an already known skill. The objective of the study is evaluate the effects of the physical practice associated with PM, on paretic MS. Subjects with unilateral stroke over 6 months, age> 18 years and who were able to hold objects will be selected. Subjects with painful conditions that affected exercise performance,> 3 spasticity by Ashworth, and cognitive deficit suggested by the Mini Mental State Examination will be excluded.

DETAILED DESCRIPTION:
There are 3 study protocols. The MP protocol 1 comprise 4 steps: 1) 5 minutes of global relaxation; 2) Video therapy, being 2 minutes / task (4 distinct tasks: stacking cubes, opposition of fingers with precision gripping, passing water from one glass to another, sequencing of bottles); 3) MP: think about the tasks assisted in the video for 5 minutes / task. 4) Physical Practice: reproduce through the motor execution, the activities assisted in the video (5 minutes / task). The MP protocol 2 was the same, changing the order: first physical practice and after MP. For the protocol 3 without PM, step 3 was suppressed, remaining the remaining steps. There were 15 sessions, 2x / week, for 1 hour. The Fugl-Meyer (FM) Scales, Ashworth Modified Scale (EMA), Functional Independence Measurement (MIF), Action Research Arm Test (ARAt), Box and block task (BBT) and Theory of mind battery (ToM) will be applied before and after the sessions, and in 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke, ischemic or hemorrhagic, for more than 6 months, age above 18 years, unilateral involvement and are able to hold objects

Exclusion Criteria:

* Painful conditions that affect the ability to perform the proposed exercises, spasticity greater than 3 by the Ashworth Scale and cognitive deficits that will be evaluated by the Mini Mental State Examination (MMSE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-06-10 (Actual); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Scale | Change from baseline sensory-motor impairmente at 8 weeks and 3 months (follow-up).
  Sensory-motor impairment of upper limb
surface electromyography | change from baseline muscle activity at 8 weeks and 3 months (follow-up)
  Short radial extensor of the carpus and superficial flexor of the fingers
Functional independence measure (FIM) | change from baseline functional independence at 8 weeks and 3 months (follow-up)
  assess the dependence of others for activities of daily living
Action Research Arm Test (ARAT) | change from baseline dexterity at 8 weeks and 3 months (follow-up)
  functional test of upper limb
Box and Block test (BBT) | change from baseline dexterity at 8 weeks and 3 months (follow-up)
  manual dexterity

SECONDARY OUTCOMES:
Movement Imagery Questionnaire-Revised second version (MIQ-RS) | change from baseline ability to imagine at 8 weeks
  evaluate the ability to imagine thick movements related to the upper and include movements referring to the ADLs.
Kinesthetic and Visual Imagery Questionnaire (KVIQ - 10) | change from baseline capacity of imagination at 8 weeks
  assessing visual and kinesthetic motor imagery
Mini-mental State Examination | baseline
  evaluation of cognition
Theory of Mind Task Battery (ToM) | change from mental function baseline at 8 weeks
  evaluation of mental function
Modified ashworth scale (MAS) | change fom baseline muscle tone at 8 weeks and 3 months (follow-up)
  evaluation of muscle tone of upper limb

CONTACTS AND LOCATIONS:
Overall Officials: Roberta O Cacho, PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Faculty of Health Science - Facisa/UFRN, Santa Cruz, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No